CLINICAL TRIAL: NCT05364996
Title: Cross-sectional Pilot Study of the Alveolar and Serum sRAGE Biomarker in Severe Asthma in Children.
Brief Title: Alveolar and Serum sRAGE in Severe Asthma in Children
Acronym: sRAGE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2021 EGRON; 2022-A00218-35 (Other: ANSM)
Record Dates: First submitted 2022-05-03; First posted 2022-05-06 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-01

CONDITIONS: Asthma in Children
Keywords: soluble receptor for advanced glycation end products; inflammation
MeSH Terms: conditions — Inflammation | interventions — Bronchoscopy; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — bronchoalveolar lavage (LBA) and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- child with severe asthma: Child eligible for bronchial endoscopy with bronchoalveolar lavage (LBA) for assessment of severe asthma. The diagnosis of asthma being established by a pneumo-pediatrician in the presence of a history of respiratory symptoms such as wheezing, shortness of breath, chest tightness and coughing variable in time and intensity, associated with a variable limitation expiratory flows.
  Interventions: Diagnostic Test: bronchial endoscopy with bronchoalveolar lavage (LBA); Diagnostic Test: Blood sampling

INTERVENTIONS:
Diagnostic Test: bronchial endoscopy with bronchoalveolar lavage (LBA) — Bronchial endoscopy under laryngeal mask and general anesthesia. BAL of saline at room temperature of 3 milliliters per kilogram limited to 20 milliliters x 3 according to recommendations
Diagnostic Test: Blood sampling — collection of 5 milliliters of blood for total white cells count, C-Reactive Protein, specific immunoglobulin E assays, serum sRAGE assay

SUMMARY:
sRAGE is a recognized marker of alveolar injury in acute respiratory distress syndrome (ARDS). More recently, it seems to be an interesting marker in asthma. It is the soluble form of the pro-inflammatory RAGE receptor overexpressed in the lungs and in particular the bronchi. It acts as a decoy to its ligands, and thus blocks the pro-inflammatory axis of RAGE.

Few studies are available in asthma, especially in children. A local study showed low levels of serum sRAGE in the context of acute bronchiolitis. The same finding emerges from the few studies available in asthma, with rates all the lower when the asthma is poorly controlled. A study carried out in the animal model in 2012 found an absence of inflammatory infiltrate, the absence of increased expression of mucin and the absence of mucus goblet cell hyperplasia within the respiratory epithelium in the absence of RAGE receptor in sensitized mice dust mites, after exposure to their allergen. One could imagine in the long term a potential therapeutic avenue by a substitution in sRAGE in this pathology.

The objective of this study is to study the ability of the alveolar sRAGE level measured on broncho-alveolar lavage for assessment, to discriminate the clinical degrees of control of severe asthma in children.

ELIGIBILITY:
Inclusion Criteria:

* severe asthma
* Weight greater than or equal to 5 kg

Exclusion Criteria:

* Current respiratory infection
* Bronchopulmonary dysplasia or prematurity < 34 weeks
* Diffuse infiltrative pneumonia
* Cystic fibrosis, primary ciliary dyskinesia
* Known immune deficiencies;
* Congenital heart disease;
* Cardiomyopathy;
* Ongoing pericarditis, myopericarditis, endocarditis;
* Chronic valvular pathology;
* Known autoimmune disease;
* Neuromuscular pathology;

Ages: 1 Day to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Child from 0 to 16 years old, eligible for bronchial endoscopy with bronchoalveolar lavage (BAL) for assessment of severe asthma. The diagnosis of asthma being established by a pneumo-pediatrician in the presence of a history of respiratory symptoms such as wheezing, shortness of breath, chest tightness and coughing variable in time and intensity, associated with a variable limitation expiratory flows.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
alveolar sRAGE level | at inclusion
  ability of the alveolar sRAGE level measured on bronchoalveolar lavage (BAL) for assessment to discriminate the clinical degrees of control of severe asthma in children

SECONDARY OUTCOMES:
plasma sRAGE level | at inclusion
  ability of the plasmatic sRAGE level measured on blood for assessment to discriminate the clinical degrees of control of severe asthma in children

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France